CLINICAL TRIAL: NCT05215561
Title: A Special Drug Use-results Survey to Evaluate the Safety and Efficacy of Subcutaneous Administration of Cosentyx in Pediatric Patients With Psoriasis Vulgaris, Psoriatic Arthritis, or Pustular Psoriasis
Brief Title: Special Drug Use-results Survey to Evaluate Safety and Efficacy of Cosentyx in Pediatric Patients With PsV, PsA, or GPP
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457L1401
Record Dates: First submitted 2022-01-19; First posted 2022-01-31 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Psoriasis Vulgaris; Psoriatic Arthritis; Pustular Psoriasis
Keywords: psoriasis vulgaris; psoriatic arthritis; pustular psoriasis; NIS; Japan; Cosentyx; pediatric
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — secukinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cosentyx: Cosentyx for Subcutaneous Injection
  Interventions: Other: Cosentyx

INTERVENTIONS:
Other: Cosentyx — There was no treatment allocation. Patients administered Cosentyx by prescription that had started before inclusion of the patient into the study were enrolled.

SUMMARY:
This was a multicenter, centrally registered observational study without a control group. This observational study was a specified drug use-results survey conducted under GPSP to collect information on safety and efficacy during the observation period (52 weeks after the start of treatment with this drug) in pediatric patients with psoriasis vulgaris, psoriatic arthritis, or pustular psoriasis who received this drug.

DETAILED DESCRIPTION:
For patients who discontinued or completed this drug before the end of the observation period, the investigator recorded adverse events that occurred within 30 days after the day following the last administration of this drug, or the day of discontinuation of the survey (the day when discontinuation of the survey was judged), whichever is later, in the CRF.

If a patient withdraw consent, information was collected during the observation period up to the date of consent withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have obtained written consent from their legally acceptable representative to cooperate in this survey before the start of treatment with this drug
* Patients aged less than 18 years at the start of treatment with this drug
* Patients newly treated with this drug for any of the following diseases: Psoriasis vulgaris, psoriatic arthritis, pustular psoriasis

Exclusion Criteria:

* Prior treatment with this drug
* Participation in an interventional study (e.g., a clinical trial) at the time of starting this drug.

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric patients who received Cosentyx
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2024-09-28 (Actual); Study Completion 2024-09-28 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse events | 52 weeks
  Incidence of SAEs was collected

SECONDARY OUTCOMES:
Subjects with psoriasis vulgaris and psoriatic arthritis: IGA mod 2011 with 0 or 1 response | Baseline, week 4, week 12, week 24 and week 52
  Investigator's Global Assessment (IGA) rating scale is:
  0 - no signs of psoriasis. Postinflammatory hyperpigmentation may be present.
  1. - Normal to pink lesions, no thickening, focal scaling absent or minimal
  2. - Pink to pale red lesions, minimal to mild thickening, and mainly fine scaling.
  3. - Clearly distinguishable erythema of dull red to bright red, clearly distinguishable to moderate thickening, moderate scaling.
  4. - Light red to dark red lesions, high thickness with hard margins, high/rough scaling covering almost all or all lesions.
Subjects with psoriasis vulgaris and psoriatic arthritis: PASI 75/90/100 response | Baseline, week 4, week 12, week 24 and week 52
  Psoriasis Area and Severity Index (PASI) 75/90 response is defined as ≥ 75%, ≥ 90% improvement (reduction) in PASI score compared to Baseline.
  PASI 100 response means no sign of body psoriasis.
All patients: Change from baseline in CDLQI | Baseline, week 4, week 12, week 24 and week 52
  Children's Dermatology Life Quality Index (CDLQI) is a global dermatology disability index designed to assess health-related quality of life in pediatric patients and consists of 10 questions about symptoms and feelings, leisure, school and holidays, personal relationships, sleep, and treatment. The total CDLQI score is the sum of 10 questions and ranges from 0 ~ 30. Higher scores indicate more impairment of health-related quality of life.
Subjects with psoriatic arthritis: Change from baseline in C-HAQ | Baseline, week 4, week 12, week 24 and week 52
  Childhood Health Assessment Questionnaire (C-HAQ) is used to assess the QOL of patients with psoriatic arthritis.
  The disability dimension consists of 20 multiple choice items concerning difficulty in performing eight common activities of daily living; dressing and grooming, arising, eating, walking, reaching, personal hygiene, gripping and other "activities". Higher scores mean worse quality of life.
Subjects with psoriatic arthritis: Change from baseline in JADAS -27 | Baseline, week 4, week 12, week 24 and week 52
  Juvenile Arthritis Disease Activity Score (JADAS) score was used to assess disease activity in patients with juvenile idiopathic arthritis including psoriatic arthritis. The investigator assessed each of the 4 components of the JADAS for patients with psoriatic arthritis (Rater's Global Assessment, Patient's or guardian's global assessment, Number of active arthritis and CRP) and record the results in the CRF. JADAS-27 is the sum of the 4 scores (0 ~ 57).
Subjects with pustular psoriasis: Change from Baseline in the Japanese Dermatological Association (JDA) Severity Index | Baseline, week 4, week 12, week 24 and week 52
  The investigator determined the severity based on the areas of erythema with pustules, areas of erythema (total), areas of edema, fever, WBC count, CRP, and serum albumin. The total score in the severity index is divided into 0 ~ 17 points (1 ~ 6 = mild, 7 ~ 10 = moderate, 11 ~ 17 = severe).
Subjects with pustular psoriasis: General improvement in GPP | Baseline, week 4, week 12, week 24 and week 52
  GPP: Generalized Pustular Psoriasis The investigator assessed the General improvement rating (Responder, partial-responder, non-responder, aggravated, indeterminate) of pustular psoriasis symptoms at each observation time point compared to the start of treatment with this drug.
Incidence of adverse events and adverse drug reactions | 52 weeks
  Incidence of AEs and ADRs was collected
Incidence of adverse events and adverse reactions included in the safety specifications | 52 weeks
  Important identified risks or important potential risks specified in the Risk Management Plan at the time of planning the surveillance were determined to be identified in the surveillance. The following items were set as the safety specifications for the surveillance:
  * Serious infections
  * Neutrophil count decreased
  * Hypersensitivity Reactions
  * inflammatory bowel disease
  * Erythroderma (exfoliative dermatitis)
  * Malignancies
  * Cardiovascular/cerebrovascular events
  * Tuberculosis
  * Events related to suicide/self-injury

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- Japan (21):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Obihiro, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Mito, Ibaraki
  - Novartis Investigative Site, Kahoku-gun, Ishikawa-ken
  - Novartis Investigative Site, Kamigyō-ku, Kyoto
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Ikoma, Nara
  - Novartis Investigative Site, Moriguchi, Osaka
  - Novartis Investigative Site, Ōsaka-sayama, Osaka
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Sumida-Ku, Tokyo
  - Novartis Investigative Site, Akita
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Wakayama

IPD SHARING:
Plan to Share IPD: No